CLINICAL TRIAL: NCT06281379
Title: Short-term Results of a Randomized Controlled Trial and Review of the Literature Complete Mesogastric Excision With D2 Lympadenectomy for Gastric Cancer: Short-term Results of a Randomized Controlled Trial and Review of the Literature
Brief Title: Complete Mesogastric Excision With D2 Lympadenectomy for Gastric Cancer:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Basaksehir City Hospital
Record Dates: First submitted 2024-02-17; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Gastric Cancer; Gastric Neoplasm; Gastric Cancer Stage
Keywords: Gastric cancer; D2 lymph node dissection; Mesogastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Study group participants: total gastrectomy+mesogastrectomy Control group: Standard total gastrectomy + D2 lymph node dissection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Total gastrectomy+mesogastrectomy
  Interventions: Procedure: Total mesogastrectomy
- Group 2 (Other): Total gastrectomy with concentional D2 lymphadenectomy
  Interventions: Procedure: Total mesogastrectomy

INTERVENTIONS:
Procedure: Total mesogastrectomy — More extended resection type with better oncological outcomes when compared to standard technique

SUMMARY:
Objective: To define complete mesogastric excision and compare our short term results for the first time in a different population.

Study design:Randomised-controlled study

Place and duration of the study: Gastroenterological Surgery Clinic,Health Sciences University,Basaksehir City Hospital,Istanbul,Turkey,from April to December 2023.

Methodology: We compared short term results of open total gastrectomy+ mesogastrectomy with standard total gastrectomy + D2 lymph node dissection at a tertiary center in terms of peroperative results, histopathological findings and postoperative short- term outcomes with review of the literature.

Conclusion: Our aim is to show that mesogastric excision is safe and has advantages over conventional D2 gastrectomy in means of not only peroperative and short-term outcomes, but also disease free survival.Our work is the first study from a different population of the world and our initial results can contribute to the literature for universalization.

DETAILED DESCRIPTION:
The curative treatment of gastrointestinal tumors is surgery referring to an en block resection of the primary tumor along with its lymphovascular drainage.Unfortunately, despite of these radical resections, published literature shows that recurrences occur in up to 38% of patients in 5 years. Morover, these rates may reach to 60% in patients with locally advanced tumor following radical surgery. However, this mesentery-based surgery is harder to apply in gastric cancer due to differences in embriyological development. In our prospective study and a review of the literature, following the descripiton of mesogastrium concept, we aimed to search and analyse former techniques and viewpoints about mesogastric excision by different surgical approaches from various countries. Later, we aimed to show our technique of mesogastrectomy, compared our short term results with limited publications from the literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histopathologically confirmed gastric adenocancer without evidence of distal metastasis and resectable tumors which have been treated with open total gastrectomy.

Exclusion Criteria:

* Patients with prior upper gastrointestinal system surgery
* Patients with neoadjuvant therapy
* Patients with peripheral organ involvement and/or distant metastasis
* Patients who underwent subtotal gastrectomy
* Patients who underwent laparoscopic and robotic operations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Postoperative outcome | Postoperative 1 week
  Complications

CONTACTS AND LOCATIONS:
Locations (1):
- Yigit Duzkoylu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 8 months

REFERENCES:
- [Background] Xie D, Gao C, Lu A, Liu L, Yu C, Hu J, Gong J. Proximal segmentation of the dorsal mesogastrium reveals new anatomical implications for laparoscopic surgery. Sci Rep. 2015 Nov 6;5:16287. doi: 10.1038/srep16287. PMID 26542081
- [Background] Girnyi S, Ekman M, Marano L, Roviello F, Polom K. Complete Mesogastric Excisions Involving Anatomically Based Concepts and Embryological-Based Surgeries: Current Knowledge and Future Challenges. Curr Oncol. 2021 Nov 22;28(6):4929-4937. doi: 10.3390/curroncol28060413. PMID 34898586
- [Background] Shinohara H, Kurahashi Y, Haruta S, Ishida Y, Sasako M. Universalization of the operative strategy by systematic mesogastric excision for stomach cancer with that for total mesorectal excision and complete mesocolic excision colorectal counterparts. Ann Gastroenterol Surg. 2017 Oct 23;2(1):28-36. doi: 10.1002/ags3.12048. eCollection 2018 Jan. PMID 29863126
- [Result] Xie D, Osaiweran H, Liu L, Wang X, Yu C, Tong Y, Hu J, Gong J. Mesogastrium: a fifth route of metastasis in gastric cancer? Med Hypotheses. 2013 Apr;80(4):498-500. doi: 10.1016/j.mehy.2012.12.020. Epub 2013 Feb 10. PMID 23403142